CLINICAL TRIAL: NCT02616328
Title: A Multicenter, Prospective, Observational, Non-Interventional Study Evaluating the Efficacy and Safety of Using Tocilizumab (TCZ) for Confirmed Rheumatoid Arthritis (RA) Patients In Clinical Practice
Brief Title: A Study of the Efficacy and Safety of Tocilizumab for Confirmed Rheumatoid Arthritis (RA) Participants in Clinical Practice
Status: Terminated | Type: Observational
Why Stopped: Planned recruitment target not reached
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29936
Record Dates: First submitted 2015-11-25; First posted 2015-11-26 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants with confirmed rheumatoid arthritis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention administered in this study

SUMMARY:
This is a single-arm, open-label, non-randomized, multicenter trial to evaluate the efficacy and safety of using tocilizumab for confirmed rheumatoid arthritis participants in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with moderate-to-severe active rheumatoid arthritis (RA) for over 3 months
* Started on tocilizumab, with or without previous history of biological treatment

Exclusion Criteria:

* Pregnant or lactating women
* Treated with an investigational drug within 30 days prior to initiation of study drug
* Having a condition that, in the opinion of the investigator, could compromise the participant's safety or interfere with the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with confirmed rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a 28-Joint Disease Activity Score (DAS28) < 2.6 at Week 24 | Week 24
Number of Participants with Adverse Events | Up to 30 months

SECONDARY OUTCOMES:
Percentage of Participants with Tender Joint Count-28 Joints (TJC28) < or = 1 at Week 12 and Week 24 | Week 12 and Week 24
Percentage of Participants with Swollen Joint Count-28 Joints (SJC28) < or = 1 at Week 12 and Week 24 | Week 12 and Week 24
Percentage of Participants with C-Reactive Protein (CRP) < or = 1mg/dL at Week 12 and Week 24 | Week 12 and Week 24
Percentage of Participants with Participant Global Health (PGH) < or = 1/10 at Week 12 and Week 24 | Week 12 and Week 24
Percentage of Participants with Clinical Disease Activity Index (CDAI) < or = 2.8 at Week 12 and Week 24 | Week 12 and Week 24
Percentage of Participants with DAS28 < or = 3.2 at Week 12 and Week 24 | Week 12 and Week 24
Percentage of Participants with CDAI < or = 10 at Week 12 and Week 24 | Week 12 and Week 24
Percentage of Participants with DAS28 < 2.6 at Week 12 | Week 12
Mean Change in DAS28 | Baseline, Week 12, and Week 24
Mean Change in CDAI | Baseline, Week 12, and Week 24
Mean Change in TJC | Baseline and Week 24
Mean Change in SJC | Baseline and Week 24
Mean Change in CRP | Baseline and Week 24
Mean Change in PGH | Baseline and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Saudi Arabia (2):
  - King Khaled Uni Hospital; Oncology, Riyadh
  - King Fahad Medical City; Gastroentrology, Riyadh